CLINICAL TRIAL: NCT02049697
Title: Absorption, Metabolism, and Excretion of 14C-JNJ-39823277 (TPI 1062) After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study to Evaluate of the Absorption, Metabolism, and Excretion of 14C-JNJ-39823277 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100588; TPI1062DEP1005 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2009-010867-17 (EudraCT Number)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Healthy; Healthy male participants; 14C-JNJ -39823277; TPI 1062; Tianeptine; Absorption; Metabolism; Excretion; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 14C-JNJ-39823277 (Experimental)
  Interventions: Drug: 14C-JNJ-39823277

INTERVENTIONS:
Drug: 14C-JNJ-39823277 — Participants will receive a single oral dose of 25 mg 14C-JNJ-39823277 as a 50-mL solution.

SUMMARY:
The purpose of this study is to investigate the absorption, metabolic pathways and excretion of JNJ-39823277 in healthy male adults after administration of a single oral dose of a 25 mg (0.5 mg/mL solution) of 14C-JNJ-39823277.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) and single-arm (group) study. The study consists of 3 phases including, the screening phase (within 3 weeks prior to the start of study medication), treatment phase (8 to 15 days), and the follow-up phase (up to 6 days after the discharge from the hospital). Approximately 6 participants will be receiving the 14C-JNJ-39823277 in the study. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored throughout the study. The total duration of study will be up to approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 20 and 30 kg/m2 (BMI will be calculated as weight [kg]/square of height [square meter])
* Had consistent bowel movement habit (approximately once per day) within 30 days before dosing
* No clinically significant laboratory and electrocardiogram abnormalities

Exclusion Criteria:

* Exposure to radiation for professional or medical reasons (exception of dental x rays and plain chest x ray) within 1 year before study medication administration
* History of or current clinically significant medical illness
* Clinically significant abnormal laboratory values, physical examination
* Positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, or barbiturates at screening and on the study medication administration

Ages: 18 Years to 56 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of 14C-JNJ-39823277 in plasma | Predose; 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours post-dose
Time of observed maximum plasma concentration (Tmax) of 14C-JNJ-39823277 | Predose; 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of 14C-JNJ-39823277 | Predose; 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours post-dose
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of 14C-JNJ-39823277 | Predose; 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours post-dose
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Elimination Half-Life Period (T1/2) of 14C-JNJ-39823277 | Predose; 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours post-dose
  T1/2 is the time measured for the plasma concentration to decrease by one-half of its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Mass Balance After an Oral Dose of 14C-JNJ-39823277 as Generated From Recovery of Total Radioactivity Excreted in Urine and Feces | Predose and up to 168 hours post-dose
Routes of 14C-JNJ-39823277 Elimination Measured Through Total Radioactivity Concentrations in Urine and Feces | Predose and up to 168 hours post-dose
Whole Blood and Plasma Partitioning of Total Radioactivity Through Measurement of Total Radioactivity Levels in Blood | Predose; post-dose 15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 120, and 168 hours
Identification of Major Metabolites in Plasma, Urine, and Feces | Predose and up to 168 hours post-dose

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerabilty | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L C.Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium